CLINICAL TRIAL: NCT03801746
Title: A Phase 1, Two-Part, Open-label Study in Healthy Adult Volunteers to Assess a Single Dose of Vadadustat as a Victim in Drug-Drug Interactions With Cyclosporine, Probenecid and Rifampin
Brief Title: Drug-Drug Interaction Study of Vadadustat With Cyclosporine, Probenecid and Rifampin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AKB-6548-CI-0029
Record Dates: First submitted 2018-12-27; First posted 2019-01-11 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Drug Interaction Potentiation
Keywords: Healthy volunteers; vadadustat; drug interactions
MeSH Terms: interventions — vadadustat; Rifampin; Probenecid; Cyclosporins

STUDY DESIGN:
Intervention Model Description: This is a 2 part study. Part 1 Arm 1 is a cross over design to assess the drug-drug interactions of cyclosporine with vadadustat. Part 1 Arm 2 is a fixed sequence design to assess the drug-drug interactions of probenecid with vadadustat. Part 2 is a crossover design to assess the drug-drug interaction of rifampin with vadadustat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat, Cyclosporine (Experimental): Part 1: Arm 1: Subjects will receive vadadustat 300 mg alone and vadadustat 300 mg in combination with oral cyclosporine 500 mg in a crossover design
  Interventions: Drug: vadadustat; Drug: Cyclosporins
- Vadadustat; Probenecid (Experimental): Part 1: Arm 2: Subjects will receive vadadustat 300 mg alone and vadadustat 300 mg in combination with oral Probenecid 500 mg Q12h in a fixed sequence design
  Interventions: Drug: vadadustat; Drug: Probenecid
- Vadadustat and Rifampin (Experimental): Part 2: Subjects will receive vadadustat 300 mg alone and vadadustat 300 mg in combination with IV rifampin 600 mg in a cross-over design
  Interventions: Drug: vadadustat; Drug: Rifampin

INTERVENTIONS:
Drug: vadadustat — Oral dose 300 mg
  Other Names: AKB 6548
Drug: Rifampin — IV Rifampin
  Arms: Vadadustat and Rifampin
Drug: Probenecid — Oral Probenecid
  Arms: Vadadustat; Probenecid
Drug: Cyclosporins — Oral Cyclosporine
  Arms: Vadadustat, Cyclosporine

SUMMARY:
This is a Phase 1, two-part, open-label study to evaluate the interaction of cyclosporine, probenecid, and rifampin as perpetrators with vadadustat (victim) in healthy male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, two-part, open-label study to evaluate the interaction of cyclosporine, probenecid, and rifampin as perpetrators with vadadustat (victim) in healthy male and female subjects. Part 1 consists of 2 arms (cyclosporine and probenecid) and Part 2 consists of 1 arm (rifampin). Twenty (20) unique subjects will be enrolled into each study arm. The PK and safety/tolerability data from Part 1 Arm 1 (cyclosporine) will determine if Part 2 (rifampin) will proceed. Subjects will be on study for up to 72 days, including a 28-day screening period, 6-10 day clinic period, and a 30-day follow-up period post last dose. Blood and/or urine samples for PK analysis will be collected at pre-defined timepoints throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female between 18 and 55 years of age, inclusive, at time of informed consent
* Body mass index between 18.0 and 30.0 kg/m2, with a minimum body weight of 45 kg for females and 50 kg for males, inclusive.

Exclusion Criteria:

* Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening; History of latent or active tuberculosis (TB).
* Positive test results for human immunodeficiency virus (HIV) antibody; Positive test results of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCVab) within 3 months prior to screening , or positive test results for human immunodeficiency virus antibody (HIVab) at Screening.
* Taking any prescription medication or over the counter multi-vitamin supplement, or any non-prescription products (including herbal-containing preparations but excluding acetaminophen) within 14 days prior to Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) of vadadustat | Up to 10 weeks
Area under plasma concentration-time curve from 0 to infinity (AUCinf) of vadadustat | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of vadadustat | Up to 10 weeks

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of vadadustat | Up to 10 weeks
Elimination rate constant (Kel) of vadadustat | Up to 10 weeks
Terminal half-life (t½) of vadadustat | Up to 10 weeks
Apparent total body clearance (CL/F) of vadadustat | Up to 10 weeks
Percent of extrapolated area under the curve from time t to infinity (%AUCextrap) of vadadustat | Up to 10 weeks
Renal clearance (CLr) of vadadustat and vadadustat 1-O-glucuronide excretion in urine for Part 1 Arm 2 (Probenecid) only | Up to 10 weeks
Cumulative amount excreted (Ae0-t) of vadadustat and vadadustat 1-O-glucuronide in urine for Part 1 Arm 2 (Probenecid) only | Up to 10 weeks
Fraction (%) of the dose excreted (Fe%0-t) for Part 1 Arm 2 (Probenecid) only of vadadustat and vadadustat 1-O-glucuronide excretion in urine | Up to 10 weeks
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) of vadadustat metabolites | Up to 10 weeks
Area under plasma concentration-time curve from 0 to infinity (AUCinf) of vadadustat metabolites | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of vadadustat metabolites | Up to 10 weeks
Reporting of treatment emergent adverse events as reported by the study subject | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Inc, Study Director — Sponsor GmbH
Locations (1):
- inVentiv Health Clinique Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided